CLINICAL TRIAL: NCT05426213
Title: A Real-World Study to Evaluate the Effectiveness and Safety of Robot-Assisted Bronchoscopy in Chinese Patients With Lung Lesions
Brief Title: A Study of Robot-Assisted Bronchoscopy in Chinese Participants With Lung Lesions
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company strategy adjustment
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDS202101; EDS202101 (Other: Auris Health, Inc.)
Record Dates: First submitted 2022-06-16; First posted 2022-06-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robot-assisted Bronchoscopy (Other): Participants with 8-50 millimeters (mm) diameter size lung lesions identified on computed tomography (CT) scan will be enrolled for robotic assisted bronchoscopy (Monarch Platform) biopsy procedure.
  Interventions: Device: Robot-assisted Bronchoscopy (Monarch Platform)

INTERVENTIONS:
Device: Robot-assisted Bronchoscopy (Monarch Platform) — Robotic assisted bronchoscopy biopsy procedures will be performed using the Monarch platform.

SUMMARY:
Robot-assisted bronchoscopy biopsy procedure will be conducted for all eligible subjects under general anesthesia status by trained investigators in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to give informed consent
* Acceptable candidate for an elective, non-emergency bronchoscopic procedure
* Lung lesions suspected of malignancy, between 8-50 millimeters (mm) in diameter size identified on thin slice (0.9-1.25 mm) computed tomography (CT) scan within 14 days, requiring bronchoscopic biopsy for diagnosis
* No more than 1 lung lesion will be targeted for robot-assisted bronchoscopy biopsy

Exclusion Criteria:

Pre-Operative

* Participants with pure ground-glass opacity lesions on pre-procedure chest CT
* Participants with the target lesion having endobronchial involvement seen on chest CT
* Medical contraindications to bronchoscopy and/or anesthesia as assessed by the investigator (such as severe cardiac arrhythmias, severe hypertension, severe cardiopulmonary dysfunction, myocardial infarction, unstable angina pectoris et cetera [etc]) precluding safe bronchoscopic procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Navigation Success Rate | Intraoperative
  Navigation success rate is defined as the percentage of successful navigation to the targeted lung lesion (lesion localization) as confirmed by radial probe endobronchial ultrasound (R-EBUS) imaging through Monarch Platform during bronchoscopy procedure.

SECONDARY OUTCOMES:
Time to R-EBUS Confirmation | Intraoperative
  Time to R-EBUS confirmation is defined by the time from the robotic bronchoscope inserted into the oropharynx to the localization of the targeted lesion confirmed by R-EBUS.
Time to the Tissue Acquisition | Intraoperative
  Time to the tissue acquisition is defined by the time the robotic bronchoscope is inserted into the oropharynx until the tissue acquisition is confirmed by the Rapid On-site evaluation (ROSE).
Total Procedure Time | Intraoperative
  Total procedure time is defined by the time the robotic bronchoscope is inserted into the oropharynx until the robotic bronchoscope is removed.
Number of Conversion to Conventional Bronchoscopic Procedure | Intraoperative
  Number of conversion to conventional bronchoscopic procedure is defined as the number of procedures converted to other diagnostic modality due to inability of the Monarch platform to complete the intended bronchoscopy.
Number of Participants with Pneumothorax Requiring Intervention | Up to 7 days post procedure
  Number of participants with pneumothorax requiring intervention (rated as greater than [>] Grade 1 according to the Common Terminology Criteria for Adverse Events [CTCAE] scale) will be reported.
Number of Participants with Device or Procedure Related Bleeding Requiring Medical Intervention | Up to 7 days post procedure
  Number of participants with device or procedure related bleeding requiring medical intervention (rated as >Grade 1 according to the CTCAE scale) will be reported.
Number of Participants with Device or Procedure Related Respiratory Failure | Up to 7 days post procedure
  Number of participants with device or procedure related respiratory failure (rated as >Grade 3 according to the CTCAE scale) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Auris Health, Inc. Clinical Trial, Study Director — Auris Health, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Zhang S, Zhao P, Zeng H, Zou X. Report of cancer incidence and mortality in China, 2010. Ann Transl Med. 2014 Jul;2(7):61. doi: 10.3978/j.issn.2305-5839.2014.04.05. PMID 25333036
- [Background] Zeng H, Chen W, Zheng R, Zhang S, Ji JS, Zou X, Xia C, Sun K, Yang Z, Li H, Wang N, Han R, Liu S, Li H, Mu H, He Y, Xu Y, Fu Z, Zhou Y, Jiang J, Yang Y, Chen J, Wei K, Fan D, Wang J, Fu F, Zhao D, Song G, Chen J, Jiang C, Zhou X, Gu X, Jin F, Li Q, Li Y, Wu T, Yan C, Dong J, Hua Z, Baade P, Bray F, Jemal A, Yu XQ, He J. Changing cancer survival in China during 2003-15: a pooled analysis of 17 population-based cancer registries. Lancet Glob Health. 2018 May;6(5):e555-e567. doi: 10.1016/S2214-109X(18)30127-X. PMID 29653628
- [Background] Cancer Stat Facts: Lung and Bronchus Cancer." National Cancer Institute, https://seer.cancer.gov/statfacts/html/lungb.html
- [Background] Kramer BS, Berg CD, Aberle DR, Prorok PC. Lung cancer screening with low-dose helical CT: results from the National Lung Screening Trial (NLST). J Med Screen. 2011;18(3):109-11. doi: 10.1258/jms.2011.011055. No abstract available. PMID 22045816
- [Background] Wood DE, Kazerooni E, Baum SL, Dransfield MT, Eapen GA, Ettinger DS, Hou L, Jackman DM, Klippenstein D, Kumar R, Lackner RP, Leard LE, Leung AN, Makani SS, Massion PP, Meyers BF, Otterson GA, Peairs K, Pipavath S, Pratt-Pozo C, Reddy C, Reid ME, Rotter AJ, Sachs PB, Schabath MB, Sequist LV, Tong BC, Travis WD, Yang SC, Gregory KM, Hughes M; National comprehension cancer network. Lung cancer screening, version 1.2015: featured updates to the NCCN guidelines. J Natl Compr Canc Netw. 2015 Jan;13(1):23-34; quiz 34. doi: 10.6004/jnccn.2015.0006. PMID 25583767
- [Background] Zhou Q, Fan Y, Wang Y, Qiao Y, Wang G, Huang Y, Wang X, Wu N, Zhang G, Zheng X, Bu H, Li Y, Wei S, Chen L, Hu C, Shi Y, Sun Y. [China National Lung Cancer Screening Guideline with Low-dose Computed Tomography (2018 version)]. Zhongguo Fei Ai Za Zhi. 2018 Feb 20;21(2):67-75. doi: 10.3779/j.issn.1009-3419.2018.02.01. Chinese. PMID 29526173
- [Background] McCarty R, Plunkett LM. Binding sites for atrial natriuretic factor (ANF) in brain: alterations in Brattleboro rats. Brain Res Bull. 1986 Dec;17(6):767-72. doi: 10.1016/0361-9230(86)90088-2. PMID 2948617
- [Background] Chen AC, Pastis NJ, Machuzak MS, Gildea TR, Simoff MJ, Gillespie CT, Mahajan AK, Oh SS, Silvestri GA. Accuracy of a Robotic Endoscopic System in Cadaver Models with Simulated Tumor Targets: ACCESS Study. Respiration. 2020;99(1):56-61. doi: 10.1159/000504181. Epub 2019 Dec 5. PMID 31805570
- [Background] Rojas-Solano JR, Ugalde-Gamboa L, Machuzak M. Robotic Bronchoscopy for Diagnosis of Suspected Lung Cancer: A Feasibility Study. J Bronchology Interv Pulmonol. 2018 Jul;25(3):168-175. doi: 10.1097/LBR.0000000000000499. PMID 29762461
- [Background] Chaddha U, Kovacs SP, Manley C, Hogarth DK, Cumbo-Nacheli G, Bhavani SV, Kumar R, Shende M, Egan JP 3rd, Murgu S. Robot-assisted bronchoscopy for pulmonary lesion diagnosis: results from the initial multicenter experience. BMC Pulm Med. 2019 Dec 11;19(1):243. doi: 10.1186/s12890-019-1010-8. PMID 31829148
- [Background] Chen AC, Pastis NJ Jr, Mahajan AK, Khandhar SJ, Simoff MJ, Machuzak MS, Cicenia J, Gildea TR, Silvestri GA. Robotic Bronchoscopy for Peripheral Pulmonary Lesions: A Multicenter Pilot and Feasibility Study (BENEFIT). Chest. 2021 Feb;159(2):845-852. doi: 10.1016/j.chest.2020.08.2047. Epub 2020 Aug 19. PMID 32822675
- [Background] Murgu S, Chen AC, Gilbert CR, Sterman DH, Pederson D, Rafeq S, Laxmanan B, Schwiers ML, Connelly J, Benz HL, Yasufuku K, Silvestri GA; TARGET Investigators. A Prospective, Multicenter Evaluation of Safety and Diagnostic Outcomes With Robotic-Assisted Bronchoscopy: Results of the Transbronchial Biopsy Assisted by Robot Guidance in the Evaluation of Tumors of the Lung (TARGET) Trial. Chest. 2025 Aug;168(2):539-555. doi: 10.1016/j.chest.2025.04.022. Epub 2025 Apr 27. PMID 40300665